CLINICAL TRIAL: NCT02386436
Title: A Phase I, Randomised, Double-blind (Sponsor Open), Placebo-Controlled Single Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2330811 in Healthy Subjects
Brief Title: A Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of GSK2330811 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201246
Record Dates: First submitted 2015-03-06; First posted 2015-03-11 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Scleroderma, Systemic
Keywords: GSK2330811; Dose Escalation; Safety; First Time in Human; Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1- GSK2330811(0.1 mg/kg) (Experimental): Subjects will be randomised to receive either 0.1 mg/kg GSK2330811 or placebo s.c single dose in a 3:1 ratio.
  Interventions: Drug: GSK2330811; Drug: Placebo
- Cohort 2- GSK2330811(0.3 mg/kg) (Experimental): Subjects will be randomised to receive either 0.3 mg/kg GSK2330811 or placebo s.c single dose in a 3:1 ratio.
  Interventions: Drug: GSK2330811; Drug: Placebo
- Cohort 3- GSK2330811(1 mg/kg) (Experimental): Subjects will be randomised to receive either 1 mg/kg GSK2330811 or placebo s.c single dose in a 3:1 ratio.
  Interventions: Drug: GSK2330811; Drug: Placebo
- Cohort 4- GSK2330811(3 mg/kg) (Experimental): Subjects will be randomised to receive either 3 mg/kg GSK2330811 or placebo s.c single dose in a 3:1 ratio.
  Interventions: Drug: GSK2330811; Drug: Placebo
- Cohort 5- GSK2330811(6 mg/kg) (Experimental): Subjects will be randomised to receive either 6 mg/kg GSK2330811 or placebo s.c single dose in a 3:1 ratio.
  Interventions: Drug: GSK2330811; Drug: Placebo

INTERVENTIONS:
Drug: GSK2330811 — GSK2330811 will be supplied as clear or opalescent, colourless, yellow to brown liquid administered as single dose s.c.
Drug: Placebo — Placebo will be supplied as Normal Saline (0.9% weight by volume [w/v] Sodium Chloride) administered as single dose s.c.

SUMMARY:
GSK2330811 is a humanised monoclonal antibody, that blocks Oncostatin M (OSM), which is being developed for the treatment of inflammatory and fibrotic diseases. This first time in human study will evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD) and immunogenicity profile of single ascending subcutaneous (s.c.) doses of GSK2330811, in healthy subjects.

This study will be a randomised, double-blind (sponsor open), placebo-controlled, single centre, single dose escalation study of s.c. administrations of GSK2330811 in healthy subjects. Approximately 40 subjects will be enrolled in the study, across 5 cohorts. Each cohort is planned to consist of 8 subjects, randomised such that 6 subjects will receive GSK2330811 and 2 subjects will receive placebo.

The starting dose for the study will be 0.1 milligram (mg)/kilogram (kg) s.c. single dose and the highest dose will be 6 mg/kg s.c. single dose. Subjects will be admitted to the clinical unit on the day prior to dosing (Day -1). On Day 1, each subject will receive a s.c. dose of GSK2330811 or placebo. Subjects will then remain as an in-patient until discharged on Day 8, after assessments have been performed. The duration of the study, including screening, is approximately 19 weeks for Cohorts 1 to 4 and 23 weeks for Cohort 5.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, vital signs and a 12-lead ECG.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Cohorts 1-4: Body weight <=100 kg and body mass index (BMI) within the range 18.5 - 29.9 kilogram per meter square (kg/m^2) (inclusive); Cohort 5: Body weight <=80 kg and BMI within the range 18.5 - 29.9 kg/m^2 (inclusive).
* Female subjects are eligible to participate if not pregnant (as confirmed by a negative serum [screening] and urine [Day -1] human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:
* Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy.
* Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until 15 weeks after dosing of study medication:
* Vasectomy with documentation of azoospermia.
* Male condom plus partner use of one of the contraceptive options as follows: Contraceptive subdermal implant that meets the Standard Operating Procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone injectable progestogen; Contraceptive vaginal ring; percutaneous contraceptive patches. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Subjects with any values for alanine aminotransferase (ALT), aspartate aminotransferase (AST), or creatinine that are above the upper limit of normal (ULN); any values for platelets or haemoglobin that are below the lower limit of normal (LLN); or any out of normal range values for white blood cells (WBC), reticulocytes, serum sodium, or serum potassium.
* Any history of gastreointestinal bleeding disorders such as peptic ulcer disease, haematemesis or other gastrointestinal bleeding.
* Subjects with medical conditions associated with increased risk of complications from bleeding.
* A history of haematological disease, such as anaemia, or acquired platelet disorders and coagulation disorders, including drug-induced thrombocytopaenia, idiopathic thrombocytopaenia or von Willebrand's disease.
* Donation of blood in excess of 500 mL within a 56 day period prior to dosing.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Clinically significant findings on ECG.
* QT duration corrected for heart rate by Fridericia's formula (QTcF) > 450 milliseconds (msec).
* History of Tuberculosis (TB) or a positive QuantiFERON®-TB Gold (trademark of Quiagen) test at screening: If the QuantiFERON®-TB Gold test is indeterminate, it can be repeated once; there must be no other clinical evidence of TB on physical examination of the subject.
* A history of carcinoma in situ and malignant disease, with the exception of basal cell carcinoma that has been completely excised prior to the study.
* Subject is unable to abstain from the use of medications known to affect platelet or clotting function, including aspirin and other nonsteroidal anti-inflammatory drugs(NSAIDs), from within five half-lives of the last dose of the platelet affecting medication prior to study day 1, until the end of study follow-up.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Smokers who would not be able to refrain from smoking whilst in the phase I unit.
* History of sensitivity to any components of the study medication, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* History of severe drug allergies, including type I hypersensitivity reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
* History of opportunistic infections within 1 year of screening or recurrent infections, as determined by the investigator.
* History of serious infection that resulted in intravenous antibiotics and/or hospitalisation within the 6 months prior to screening.
* Active bacterial infection, viral infection, or fever >38 degree centigrade within 14 days prior to Day 1.
* A history of frequent reactivation of herpes simplex.
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening or within 3 months prior to dosing study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody at screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical or four new biological entities within 12 months prior to the first dosing day.
* Subject is unable to abstain from travelling to regions of high endemic infection, as determined by the investigator, for the duration of the study.
* Subject is unable to abstain from being immunised with live-attenuated vaccines for 4 weeks prior to day 1, until the end of follow up.
* Subject is unable to refrain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study.
* For cohorts including suction blisters (Cohorts 3-5 only): Presence of skin abnormalities that would either interfere with study procedures (for example; tattoos, naevi, sun burn/sun bed use within 7 days) or increase the risk to the subject (for example: history of keloids, skin allergy, hypersensitivity or contact dermatitis, including previous reactions to dressings to be used in the study), as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-04-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by number of subjects with adverse event (AEs) and serious adverse events (SAEs) | From Day 1 up to Day 105 (For Cohort 5 up to Day 133)
Safety and tolerability as assessed by composite of clinical laboratory tests: clinical chemistry, hematology and urinalysis | From Day 1 up to Day 105(For Cohort 5 up to Day 133)
  Clinical laboratory tests will include clinical chemistry, hematology and urinalysis.
Safety and tolerability as assessed by composite of vital signs assessment: blood pressure, heart rate and temperature | From Day 1 up to Day 105 (For Cohort 5 up to Day 133)
  Vital signs assessment including systolic and diastolic blood pressure, heart rate and body temperature.
Safety as assessed by electrocardiogram (ECG) measurements | From Day 1 up to Day 105
  ECGs will be measured in the semi-supine position. Triplicate 12-lead ECGs will be recorded at screening, Day 1 pre-dose and Day 5 and single 12-lead ECGs at all other time points.

SECONDARY OUTCOMES:
Composite PK parameters including Cmax, AUC, t1/2 and Vss/F after single s.c. doses of GSK2330811 in healthy subjects | Samples will be collected at pre-dose and at 8 hours post dose on Day 1 and single sample on Day 2, Day 3, Day 5, Day 7, Day 10, Day 14, Day 21, Day 28, Day 42, Day 56, Day 84, Day 105 and Day 133
  PK parameters will include maximum observed concentration (Cmax), area under concentration-time curve (AUC), terminal phase half-life (t1/2), and Steady State Volume of Distribution / Bioavailability (Vss/F)
Plasma concentrations of GSK2330811 | Samples will be collected at pre-dose, and at 8 hours post dose on Day 1 and single sample on Day 2, Day 3, Day 5, Day 7, Day 10, Day 14, Day 21, Day 28, Day 42, Day 56, Day 84, Day 105 and Day 133
  Plasma concentration of GSK2330811 will be determined from blood samples collected at various time points indicated in timeframe.
Incidence, specificity and titers of anti-GSK2330811 antibodies | Samples will be collected at pre-dose, Day 14, Day 28 and Day 105.
  Serum samples from 4 millilitre (mL) of whole blood will be collected to evaluate incidence, specificity and titers of anti-GSK2330811 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 201246 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201246?search=study&search_terms=201246#rs